CLINICAL TRIAL: NCT04020042
Title: Timely Epidural Placement Using Handheld Ultrasound Device vs. Traditional Landmark Palpation in Parturients With Various Body Mass Indices (BMI): A Prospective Randomized Clinical Trial
Brief Title: Epidural Placement Using Handheld Ultrasound Device vs. Traditional Landmark Palpation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Manpower issues
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Weike Tao, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU-2019-0571
Record Dates: First submitted 2019-07-12; First posted 2019-07-15 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound imaging guidance (Experimental): Determination of epidural needle site by using ultrasound guidance
  Interventions: Other: Ultrasound image guidance
- Traditional landmark palpation (Active Comparator): Depermination of epidural needle site by using traditional landmark method
  Interventions: Other: Landmark palpation

INTERVENTIONS:
Other: Ultrasound image guidance — Epidural landmarks will be determined with using ultrasound image
  Arms: Ultrasound imaging guidance
Other: Landmark palpation — Epidural landmarks will be determined with palpation
  Other Names: Determination of epidural lanmakrks with palpation
  Arms: Traditional landmark palpation

SUMMARY:
Ultrasound is widely in uses for vascular, nerve block and sometimes neuraxial block. The purpose of the study is to evaluate the impact of a handheld ultrasound device on the time to complete labor epidural placement and success rate of epidural analgesia in parturients with a wide range of body mass indexes (BMIs).

A handheld ultrasound device (Accuro, Rhivanna Medical, Charlottesville, VA) may eliminate the time for equipment setup due to its portability and instant power-up. In addition, it provides a simulated diagram to aid in identifying bone and lumbar spaces. These unique features may be helpful in laboring women with a particular BMI range. We aim to define the usefulness of guidance with a handheld ultrasound in completing labor epidural analgesia in various BMIs.

The primary outcome: The time needed to complete epidural placements.

Secondary outcomes:

* The number of needle insertion attempts,
* The rate of success measured by the need to replacements during the labor course for vaginal or cesarean delivery.

DETAILED DESCRIPTION:
This randomized prospective clinical trial aims to evaluate timing savings in performing labor epidural analgesia and the success rate of labor analgesia with and without the guidance of a handheld ultrasound device in various BMI groups.

In routine clinical setting, patients admitted to clinic and evaluated labor condition. If patient in active labor and request epidural for labor pain, the standard care team inform obstetric anesthesia epidural team by using pager. Standard of care anesthesia epidural team perform preoperative evaluation and placed the catheter.

The patients in active labor will receive labor epidural analgesia, regardless of the study participation. There is no changes epidural local anesthetic type and doses. The research intervention is only placing hand-hold ultrasound to the back of the patient and see the land mark visually before the epidural catheter placement. The remaining catheter placement is the same as the control group.

Study Procedures:

A Total of 300 eligible parturients will be randomly assigned to one of the two groups either the ultrasound imaging guidance or the traditional landmark palpation group for labor epidural needle placement. The research intervention is simply placing a hand-held ultrasound device on the back of the patient and insert the epidural needle with ultrasound image guidance.

Parturient will receive epidural catheter regardless of the study participation. In the traditional landmark method, anesthetist palpates the structure to determine the site of the initial needle insertion site. The needle will be protruded as in usual standard practice. Anesthetist may remove and insert needle again until feeling epidural space. When anesthetist determine the tip of the needle is in the epidural space, the epidural catheter will be protruded through the needle.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Parturient in active labor and desires labor epidural for pain relief.
* American Society of Anesthesiologists (ASA) Class I, 2 and 3 parturients, which include normal parturients
* Parturients with morbidities (including obesity) that are not life-threatening,
* Parturient BMI ≥ 25

Exclusion Criteria:

* History of scoliosis or back surgery
* Patient refusal
* Patient with elevated intracranial pressure
* Any patient with a contraindication for placement of epidural anesthesia, including infection at needle insertion site, or coagulopathy.
* ASA Class 4

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
The time needed to complete epidural placements | Within 10 minutes during epidural needle placement
  The number of removal and insertion of the epidural needle until feeling epidural space.

SECONDARY OUTCOMES:
The number of needle insertion attempts | Within 10 minutes during epidural needle placement
  The epidural needle insertion attempts

CONTACTS AND LOCATIONS:
Overall Officials: Seema Dave, MPH, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health Hospital System, Dallas, Texas, United States